CLINICAL TRIAL: NCT05339178
Title: Evaluation of the Quality of Life of Periodontitis Patients Visiting Supportive Periodontal Therapy - A Prospective Study
Brief Title: Quality of Life of Periodontitis Patients Visiting Supportive Periodontal Therapy
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Kristina Bertl, Principal Investigator, Medical University of Vienna
Other Study IDs: 1398/2021
Record Dates: First submitted 2022-04-08; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Quality of Life; Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present prospective study aims to assess the QoL of periodontitis patients during supportive treatment and to relate it to periodontal health (clinical and radiographic data) and treatment stability. Follow-ups after the first cross-sectional assessment are planned after approximately 2.5, 5, 7.5, and 10 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients returning for supportive therapy on a regular basis after active periodontal treatment will be asked for participation if they are in supportive therapy for at least 1 year.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: periodontitis patients undergoing supportive treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
disease specific OHRQoL (ParoQoL) | at baseline
disease specific OHRQoL (ParoQoL) | after 2.5 years
disease specific OHRQoL (ParoQoL) | after 5 years
disease specific OHRQoL (ParoQoL) | after 7.5 years
disease specific OHRQoL (ParoQoL) | after 10 years

SECONDARY OUTCOMES:
Oral Health Impact Profile (OHIP) | at baseline
perceived stress scale (PSS) | at baseline
overall health status of the patients (EQ5D-5L) | at baseline
Oral Health Impact Profile (OHIP) | after 2.5 years
perceived stress scale (PSS) | after 2.5 years
overall health status of the patients (EQ5D-5L) | after 2.5 years
Oral Health Impact Profile (OHIP) | after 5 years
perceived stress scale (PSS) | after 5 years
overall health status of the patients (EQ5D-5L) | after 5 years
Oral Health Impact Profile (OHIP) | after 7.5 years
perceived stress scale (PSS) | after 7.5 years
overall health status of the patients (EQ5D-5L) | after 7.5 years
Oral Health Impact Profile (OHIP) | after 10 years
perceived stress scale (PSS) | after 10 years
overall health status of the patients (EQ5D-5L) | after 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Oral Surgery, School of Dentistry, Medical University of Vienna, Vienna, Austria